CLINICAL TRIAL: NCT05124951
Title: The Efficacy of Whole-ventricle Irradiation Plus Primary Boost in Patients With Localized Basal Ganglia Germ Cell Tumors: Prospective Phase II Study
Brief Title: The Efficacy of WVI in Patients With Localized Basal Ganglia Intracranial Germ Cell Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Tao Jiang, Principal investigator, Beijing Tiantan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-IGCT-001
Record Dates: First submitted 2021-10-13; First posted 2021-11-18 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Intracranial Germ Cell CNS Tumor, Childhood
Keywords: intracranial germ cell tumors; basal ganglia; radiotherapy; target volume; quality of life
MeSH Terms: interventions — EC regimen; Ifosfamide; PE regimen; Second-Look Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- iGCTS (Experimental): Stratum I (Germinoma) Patients who achieved complete response after induction chemotherapy will receive WVI 2400cGy/15f plus primary boost 640cGy/4f.
  Stratum II (NGGCTs) At the time of response evaluation before radiotherapy, those with complete response or residue disease <1.5cm will receive WVI 3060cGy/17f plus primary boost 2340cGy/13f.
  Interventions: Radiation: Whole-ventricle irradiation; Drug: Carboplatin/etoposide; Drug: Ifosfamide/cisplatin/etoposide; Procedure: Second-look surgery

INTERVENTIONS:
Radiation: Whole-ventricle irradiation — Whole-ventricle irradiation will be applied in patients with localized basal ganglia germ cell tumors after induction chemotherapy
Drug: Carboplatin/etoposide — Carboplatin/etoposide regimen is applied as induction chemotherapy in patients with basal ganglia germinoma
Drug: Ifosfamide/cisplatin/etoposide — Ifosfamide/cisplatin/etoposide regimen is applied as induction chemotherapy in patients with basal ganglia non-germinomatous germ cell tumors.
Procedure: Second-look surgery — Second-look surgery would be applied to patients who presented residue disease after induction chemotherapy.

SUMMARY:
Primary endpoint

1. three-year disease-free survival of patients with localized basal ganglia germ cell tumors receiving whole-ventricle irradiation
2. Health-related quality of life measured by PedsQL 4.0 and SF-36

Second endpoint

1. three-year overall survival of patients with localized basal ganglia germ cell tumors receiving whole-ventricle irradiation
2. Adverse effects of chemoradiotherapy measured by NCI CTCAE 5.0

DETAILED DESCRIPTION:
Intracranial germ cell tumors originating from the basal ganglia area are rare, accounting for less than 20% of patients. Radiotherapy played a vital role in the treatment of this malignancy. However, the optimal target volume is still undetermined.

Our study regarding relapse patterns of different radiation volumes showed that the ventricular system and ipsilateral frontal lobe were at risk of relapse after focal radiotherapy. Although craniospinal irradiation (CSI) and whole-brain irradiation (WBI) could significantly reduce the relapse in the above areas, the adverse effect on the quality of life is still a concern. As a result, the investigators proposed whole-ventricular irradiation (WVI) in patients with localized basal ganglia germ cell tumors. In order to evaluate its efficacy and safety, the investigators designed this phase II study.

ELIGIBILITY:
Stratum I: germinoma

Inclusion Criteria:

* 3 years ≤ age ≤ 30 years
* Newly diagnosed
* Unilateral basal ganglia/thalamus lesion
* Germinoma：Histologically confirmed; and/or serum and/or CSF beta-HCG elevation (≤50IU/L); AFP negative
* No radiological evidence of additional lesions in the CNS
* Negative CSF cytology test
* Adequate organ function
* Written informed consent

Exclusion Criteria:

* Bilateral basal ganglia/ thalamus lesions
* Synchronous pineal or sellar/suprasellar lesion
* Diabetes insipidus
* With extracranial lesion(s)
* Serum/CSF β-HCG >50IU/L without histology
* Mature teratoma with normal tumor markers
* Inadequate organ function
* Poor compliance

Stratum II: non-germinomatous germ cell tumors

Inclusion Criteria:

* 3 years ≤ age ≤ 30 years
* Newly diagnosed
* Unilateral basal ganglia/thalamus lesion
* NGGCTs: Histologically confirmed; and/or serum and/or CSF AFP elevation; beta-HCG≥500IU/L
* No radiological evidence of additional lesions in the CNS
* Negative CSF cytology test
* Adequate organ function
* Written informed consent

Exclusion Criteria:

* Bilateral basal ganglia/ thalamus lesions
* Synchronous pineal or sellar/suprasellar lesion
* Diabetes insipitus
* With extracranial lesion(s)
* 50IU/L<serum/CSF β-HCG <500IU/L without histology
* Mature teratoma with normal AFP and β-HCG <500IU/L
* Inadequate organ function
* Poor compliance

Ages: 3 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
3-year event-free survival | From the enrollment to the event (relapse or death of any cause), approximately 3 years. The patients will receive long-term follow-up including MRI and serum tumor markers examination every 3 months until 36 months.
  Event-free survival (DFS) is calculated from the date of enrollment to the date of an event (relapse or death of any cause).
Change of score of the QoL questionnaire (PedsQL 4.0 : Pediatric Quality of Life Inventory Version 4.0 Generic Core Scales, Chinese edition) | Score will be obtained at baseline, 6 months posttreatment, yearly through 3 years posttreatment
  The PedsQL 4.0 Generic Core Scale contains 23 items that measures physical (eight items), emotional (five items), social (five items), and school (five items) functions. The Scale comprises parallel patient self-report and parent proxy-report formats. The items are reverse-scored and trans- formed to a 0-100 scale according to the instructions, and higher scores indicate a better HRQOL. (age ≤18 years)
Change of score of the QoL questionnaire (Short form-36) | Evaluation will be conducted at baseline, 6 months posttreatment, yearly through 3 years posttreatment
  Altogether, 36 questions with standardized response choices were organized into eight scales, including physical functioning (PF), role limitations as a result of physical health problems (RP), body pain (BP), general health perceptions (GH), vitality (VT), social functioning (SF), role limitations as a result of emotional problems (RE), and general mental health (MH). Additionally, reported health transition (HT) was used to evaluate general health changes during the previous year. The raw scores were converted to a 0-100 scale according to the instructions, and higher scores indicated a better HRQOL. Physical component score (PCS) and mental component score (MCS) were also calculated. (Age >15 years)
Change of score of Chinese Wechsler Intelligence Scale for Children | Score will be obtained at baseline, 6 months posttreatment, yearly through 3 years posttreatment
  The intelligence of the child was tested by the China-Wechsler Intelligence Scale for Children (C-WISC), which was revised by Gong and Cai at Hunan Medical University. The C-WISC consists of 11 individual tests that include six verbal tests [Information (I), Comprehend (C), Sorting (S), Arithmetic (A), Vocabulary (V), and Digit symbol (D)] and five performance tests [Picture Completing (PC), Picture Arrangement (PA), Block Pattern (BP), Object Assembly (OA), and Coding (CD)]. Based on individual testing, vocabulary scores (V), procedure scores (P), and full scores (F) were obtained. Furthermore, the VIQ, PIQ, and full intelligence quotient (FIQ) were calculated progressively .

SECONDARY OUTCOMES:
3-year overall survival | From the enrollment to the death of any cause or last follow-up, approximately 3 years.The patients will receive long-term follow-up including MRI and serum tumor markers examination every 3 months until 36 months.
  Overall survival is determined from the date of diagnosis to the date of death of any cause or the last follow-up visit
Short-term adverse effects of treatments | From the beginning to the completion of chemoradiotherapy, approximately 6 months. Grade 3/4 toxicities will be documented
  NCI CTCAE 5.0 will be used for adverse effects evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Tao Jiang, MD, PhD, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, China